CLINICAL TRIAL: NCT07015983
Title: A Phase 2, Multicenter, Open-Label Study of CC-97540 (BMS-986353), CD19-Targeted NEX-T CAR T Cells, in Participants With Active SLE (Including Lupus Nephritis) With Inadequate Response to Glucocorticoids and at Least 2 Immunosuppressants (Breakfree-SLE)
Brief Title: A Study of CC-97540 (BMS-986353 or Zola-cel), CD19-Targeted NEX-T CAR T Cells, in Participants With Active SLE Despite Immunosuppressants (Breakfree-SLE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA061-1011; 2024-519278-37 (Other: EU CTR)
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Nephritis
Keywords: Lupus; SLE; LN; CAR T; Cell Therapy; CD19 CAR T; CD19; CD19 NEX-T; CD19 NEXT; CD19 NEX T; Zola-cel; Zolacabtagene autoleucel
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-97540 (Experimental)
  Interventions: Drug: CC-97540; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CC-97540 — Specified dose on specified days
  Other Names: BMS-986353; Zola-cel; Zolacabtagene autoleucel
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and drug levels of CC-97540 in participants with active systemic lupus erythematosus (SLE) including lupus nephritis with inadequate response to glucocorticoids and at least 2 immunosuppressants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet EULAR/ACR 2019 criteria for SLE.
* Participants must have an inadequate response to appropriate doses of glucocorticoids and ≥ 2 immunosuppressant therapies, used for at least 3 months.
* Participants must have active disease when signing ICF.

Exclusion Criteria:

* Participants must not have other diseases, conditions, or treatments that may confound interpretation of the effects of CC-97540 in SLE.
* Uncontrolled or clinically significant cardiovascular conditions or CNS pathology participants must not have prior history of malignancies or lymphoproliferative disease, unless the participant has been free of the disease for ≥ 2 years, except for some non-invasive malignancies.
* IOCBP who are pregnant, nursing, or breastfeeding, or who intend to become pregnant during participation in the study.
* Participants must not have prior treatment with CAR T cell therapy, genetically modified T cell therapy, stem cell transplant or organ transplant.
* Participants must not have received live vaccines within 6 weeks before LDC (lymphodepleting chemotherapy) administration.
* Participant must not have inadequate organ function.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2028-05-17 (Estimated); Study Completion 2032-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving drug-free Definition of Remission in Systemic Lupus Erythematosus (DORIS) remission | At month 6

SECONDARY OUTCOMES:
Complete renal response (CRR) for participants with baseline lupus nephritis (LN) | Up to Month 60
Participants with drug-free DORIS remission | Up to month 60
CRR for participants with baseline LN | Up to month 60
Modified CRR for participants with baseline LN | Up to month 60
Number of participants achieving Lupus Low Disease Activity State (LLDAS) with baseline Systemic Lupus Erythematosus Disease Activity Questionnaire (SLEDAI) ≥6 | Up to month 60
Number of participants achieving SLE Responder Index (SRI) - 4 with baseline SLEDAI ≥6 | Up to month 60
Number of participants with flares as assessed by SLEDAI flare index | Up to month 60
Severity of participants with flares as assessed by SLEDAI flare index | Up to month 60
Change from baseline in proteinuria | Up to month 60
Change from baseline in estimated glomerular filtration rate (eGFR) | Up to month 60
Change from baseline in Systemic Lupus International Collaborating Clinics (SLICC)/ACR (American College of Rheumatology) damage index | Up to month 60
Percentage of participants achieving maintenance of drug-free DORIS remission | Up to month 60
Percentage of participants achieving maintenance of LLDAS | Up to month 60
Percentage of participants achieving maintenance of SRI-4 | Up to month 60
Time from first response to loss of response for drug-free DORIS remission | Up to month 60
Time from first response to loss of response for LLDAS | Up to month 60
Time from first response to loss of response for SRI-4 | Up to month 60
Time from baseline to first drug-free DORIS remission | Up to month 60
Time from baseline to LLDAS | Up to month 60
Time from baseline to SRI-4 | Up to month 60
Duration of drug-free status | Up to month 60
Percentage of participants achieving DORIS remission regardless of drug-free status | Up to month 60
Glucocorticoid used post-infusion for SLE treatment | Up to month 60
Change of serum autoantibodies from baseline | Up to month 60
Change in complement factor (C3 and C4) levels from baseline | Up to month 60
Change from baseline in patient reported outcomes (PRO) as assessed by FACIT-Fatigue | Up to month 60
Change from baseline in PRO as assessed by SF 36 v2 Acute | Up to month 60
Change from baseline in PRO as assessed by EQ-5D-5L | Up to month 60
Change from baseline in PRO as assessed by Patient Global Impression of Severity (PGI-S) Pain | Up to month 60
Change from baseline in PRO as assessed by PGI-S Fatigue | Up to month 60
Patient Global Impression of Change (PGI-C) Pain | Up to month 60
PGI-C Fatigue | Up to month 60
Number of participants with Adverse Events (AEs) | Up to month 60
Number of participants with serious AEs (SAEs) | Up to month 60
Number of participants with AESIs (AEs of Special Interest) | Up to month 60
Number of participants with clinically significant laboratory abnormalities | Up to month 60

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (93):
- United States (39):
  - Local Institution - 0009, Birmingham, Alabama
  - Local Institution - 0080, Scottsdale, Arizona
  - Local Institution - 0038, Los Angeles, California
  - Local Institution - 0051, Los Angeles, California
  - Local Institution - 0093, Newport Beach, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Local Institution - 0097, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Local Institution - 0073, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - USF Health, Tampa, Florida
  - Florida Medical Clinic Orlando Health, Zephyrhills, Florida
  - Local Institution - 0076, Athens, Georgia
  - Local Institution - 0078, Atlanta, Georgia
  - Local Institution - 0079, Atlanta, Georgia
  - Local Institution - 0074, Honolulu, Hawaii
  - Local Institution - 0086, Baton Rouge, Louisiana
  - Local Institution - 0094, Boston, Massachusetts
  - Local Institution - 0052, Boston, Massachusetts
  - Local Institution - 0096, Ann Arbor, Michigan
  - Local Institution - 0011, Rochester, Minnesota
  - Atlantic Health System Overlook Medical Center, Summit, New Jersey
  - Local Institution - 0082, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Local Institution - 0005, New York, New York
  - Local Institution - 0095, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Local Institution - 0010, Chapel Hill, North Carolina
  - Local Institution - 0065, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 0041, Oklahoma City, Oklahoma
  - Local Institution - 0083, Philadelphia, Pennsylvania
  - Local Institution - 0092, Memphis, Tennessee
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- Argentina (4):
  - Local Institution - 0016, ABB, Buenos Aires F.D.
  - Local Institution - 0017, ABB, Buenos Aires F.D.
  - Local Institution - 0023, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0077, Córdoba
- Austria (2):
  - Medizinische Universität Wien, Vienna, Vienna
  - Uniklinikum Salzburg, Salzburg
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium
- Brazil (3):
  - Local Institution - 0058, São Paulo, São Paulo
  - Local Institution - 0021, São Paulo
  - Local Institution - 0022, São Paulo
- Canada (2):
  - Local Institution - 0048, Vancouver, British Columbia
  - Local Institution - 0045, Toronto, Ontario
- Denmark (2):
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Local Institution - 0047, Copenhagen
- France (4):
  - Local Institution - 0081, Toulouse, Haute-Garonne
  - CHU Montpellier Lapeyronie Hospital, Montpellier, Hérault
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
  - Pitie Salpetriere University Hospital, Paris, Île-de-France Region
- Germany (6):
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité - Universitaetsmedizin Berlin - Campus Bejnamin Franklin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Erlangen, Erlangen
  - Local Institution - 0084, Herne
- Israel (2):
  - Local Institution - 0043, Ramat Gan, Central District
  - Local Institution - 0042, Jerusalem
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Rome, Lazio
  - Local Institution - 0032, Milan, Milano
  - Local Institution - 0044, Rome, Roma
  - Local Institution - 0070, Pisa, Tuscany
- Japan (8):
  - Local Institution - 0055, Sapporo, Hokkaido
  - Local Institution - 0072, Yokohama, Kanagawa
  - Local Institution - 0068, Bunkyo-ku, Tokyo
  - Local Institution - 0069, Shinjuku-ku, Tokyo
  - Local Institution - 0067, Chiba
  - Local Institution - 0054, Fukuoka
  - Local Institution - 0063, Okayama
  - Local Institution - 0053, Osaka
- Local Institution - 0046, Amsterdam, North Holland, Netherlands
- Poland (3):
  - Szpital Specjalistyczny nr 1 w Bytomiu, Bytom, Silesian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach, Gliwice, Silesian Voivodeship
  - Local Institution - 0034, Lodz, Łódź Voivodeship
- Local Institution - 0013, Lisbon, Lisbon District, Portugal
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Local Institution - 0088, Donostia / San Sebastian, Gipuzkoa
  - Local Institution - 0087, Madrid
  - H.R.U Málaga - Hospital General, Málaga
- United Kingdom (6):
  - Local Institution - 0061, London, London, City of
  - University College London Hospital, London, London, City of
  - King's College Hospital, London, London, City of
  - Local Institution - 0057, London, London, City of
  - Local Institution - 0090, Metropolitan Borough of Wirral, Merseyside
  - Local Institution - 0091, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07015983.html